CLINICAL TRIAL: NCT01052324
Title: The Effect Site Concentration of Remifentanil for Conscious Sedation During Awake Nasotracheal Fiberoptic Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Yuen Hee Shim, MD, PhD, Professor of Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Reseach Institute, Yonsei University College of Medicine, Seoul, Republic of Korea
Purpose: Prevention
Other Study IDs: 4-2009-0609
Record Dates: First submitted 2010-01-11; First posted 2010-01-20 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Cervical Disc Herniation; Cervical Spinal Stenosis; Cervical Spine Damage
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Remifentanil — After topical airway anesthesia with 10 % lidocaine in nostril and oropharyx, 1.5~2.0 mg of IV midazolam is injected. Awake nasotracheal fiberoptic intubation is performed with target-controlled infusion of remifentanil. Initial effect site concentration is 3.0 ng/ml. Smooth intubation is defined as absence of persistent cough with head elevation and defensive movement of extremities. In case of smooth intubation, effect site concentration is decreased by 0.5 ng/ml for the subsequent case. If intubation is not smooth, effect site concentration is increased by 0.5 ng/ml for the subsequent case. EC50 of remifentanil is determined using Dixon's up-and-down method.

SUMMARY:
Remifentanil provides analgesia, suppresses airway reflex, has little effect on cognitive function. It can be used for conscious sedation during awake nasotracheal fiberoptic intubation. Target-controlled infusion is more reliable technique for maintaining optimal infusion rate than manual controlled infusion. The aim of this study is to determine the effect site concentration of remifentanil for successful conscious sedation during awake nasotracheal fiberoptic intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cervical spine surgery
* Age 20-65
* American Society of Anesthesiologists physical status classification I or II

Exclusion Criteria:

* Patients' refusal
* allergy to any drug used
* unable to cooperate
* Severe hepatic or renal disease
* coagulation disorder
* chronic use of opioids or sedatives
* increase risk of pulmonary aspiration.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
EC50 of remifentanil for preventing persistent cough and defensive movement using Dixon's up-and-down method

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Hee Shim, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea